CLINICAL TRIAL: NCT05827575
Title: Transcutaneous Auricular Vagal Nerve Stimulation for Functional Dyspepsia With Sleep Disturbances: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022006
Record Dates: First submitted 2023-01-16; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Functional Dyspepsia; Sleep Disturbances
Keywords: Transcutaneous Auricular Vagal Nerve Stimulation; Functional Dyspepsia; Sleep Disturbances
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS (Experimental): selected cavum conchae of the two ears for 25hz electrical stimulation
  Interventions: Device: Transcutaneous Auricular Vagal Nerve Stimulation
- sham-taVNS (Sham Comparator): selected scapha of the two ears for 25hz electrical stimulation
  Interventions: Device: Transcutaneous Auricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagal Nerve Stimulation — stimulation on both ear within different area for 4 weeks；parameter：2s on，3s off,0.5ms，25hz

SUMMARY:
Functional dyspepsia(FD) is most common in functional gastrointestinal disorders whose rick factors include sleep disturbances. The medication treatment for functional dyspepsia with sleep disturbances has disadvantages such as addiction and withdrawal symptoms. Transcutaneous auricular vagal nerve stimulation(taVNS) is a new therapeutic method to improve dyspepsia and sleep. Study on taSNS for FD with sleep disturbances has not yet been explored.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is most common in functional gastrointestinal disorders whose risk factors include sleep disturbances. The medication treatment for FD with sleep disturbances has disadvantages such as addiction and withdrawal symptoms. Transcutaneous auricular vagal nerve stimulation (taVNS) is a new therapeutic method to improve dyspepsia and sleep. The study on taVNS for FD with sleep disturbances has not yet been explored.60 participants who have FD and sleep disturbances are recruited from the department of the Second Affiliated Hospital of Xi'an Jiaotong University. Inclusion criteria follows: meeting the ROME IV diagnostic criteria of FD; Pittsburgh Sleep Quality Index(PSQI)>7; aged 18-65 years old; not taking related drugs in past one month; from March 2022 to June 2023; sign informed consent. All patients were randomly divided into 2 groups and respectively treated with taVNS and sham-taVNS for four weeks. PSQI, Nepean dyspepsia index (NDI), electrogastrogram (ECG), nutrient drinking satiety test, Hamilton Anxiety and Depression Scale, heart rate variability (HRV) and serum melatonin (MLT) were recorded at baseline and after 4-week treatment. The effect and mechanism of taVNS for FD with sleep disturbances were investigated by comparing the indexes before and after treatment of taVNS and sham-taVNS groups. The study was proved by the medical ethics committee of the Second Affiliated Hospital of Xi'an Jiaotong University.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Functional bloating/distension with Rome IV;
2. Pittsburgh Sleep Quality Index(PSQI)>7;
3. Aged 18-65 years old；

Exclusion Criteria:

1. Have taken drugs that may affect gastrointestinal motility and sleep in the past two week;
2. The history of gastrointestinal surgery;
3. With severe heart, liver and kidney diseases;

5.Pregnant and breastfeeding women; 6.Skin allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Dyspepsia score | after 4 weeks taVNS treatment
  Nepean Dyspepsia Index：the symptom severity score and life quality score
Sleep score | after 4 weeks taVNS treatment
  Pittsburgh Sleep Quality Index
Hamilton Anxiety and Depression Scale score | after 4 weeks taVNS treatment
  Score of Hamilton Anxiety and Depression Scale
Gastric slow waves in electrogastrograph | after 4 weeks taVNS treatment
  The percentage of the normal gastric slow waves in fasting, fed states and the post-preprandial EGG power ratio
The threshold volume(TV)and maximal volume（MV） | after 4 weeks taVNS treatment
  Nutrient drinking satiety test: drink [100 g milk powder, 50 g chocolate powder (Cola Coa, Idilia Foods), and 1,120 mL water (0.6 Cal/mL, fat:19%, protein: 18%, carbohydrate: 63%)] at a speed of 60mL/min until reaching the threshold volume(TV)and maximal volume（MV).
Heart rate variability（HRV） | after 4 weeks taVNS treatment
  Assessment of autonomic function with heart rate variability
Serum melatonin (MLT) level | after 4 weeks taVNS treatment
  test the level of serum melatonin

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China